CLINICAL TRIAL: NCT00836524
Title: "Kan IUGR og præeclampsi Forudsiges ud Fra YKL-40 målt i Serum?" "Metoder Til at Vurdere om Den Gravide Har Risiko for at Udvikle Svangerskabsforgiftning og/Eller væksthæmning Hos Fosteret".
Brief Title: Is Serum YKL-40 Capable of Predicting Intrauterine Growth Restriction (IUGR) and Preeclampsia?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: Region Zealand (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Dorte Nymark Brask, MD, phd student, Zealand University Hospital
Other Study IDs: SJ-55
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Intrauterine Growth Restriction; Preeclampsia
Keywords: IUGR; Preeclampsia; ultrasound; YKL-40
MeSH Terms: conditions — Fetal Growth Retardation; Pre-Eclampsia | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloodsamples will be collected as well as placenta tissue for histology.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Pregnant women are included when they attend nuchal transcluency examination and will during their pregnancy be examined 4 times with ultrasound
  Interventions: Procedure: ultrasound

INTERVENTIONS:
Procedure: ultrasound — 4 ultrasound examinations during pregnancy and every time a blood sample is colletted. blood sample from the mother and the umbilical cord is collected as well

SUMMARY:
Objective: To investigate the role of maternal serum YKL-40 and uterine artery doppler, at gestational age 12, 20, 25 and 32 weeks, and the relation to preeclampsia and intrauterine growth restriction. The serum marker YKL-40 is related to conditions involving inflammation, infection, tissue remodeling, fibrosis and cancer. IUGR and preeclampsia are known to be related to inflammation and tissue remodeling.

Methods: women attending screening for downs syndrome is scanned with uterine artery doppler and delivered blood samples at GA 12, 20, 25 and 32 respectively. When pregnancy outcome is registered by medical records blood samples are retrieved and analyzed for serum YKL-40. Serum YKL-40 are correlated to the presence of bilateral notching, preeclampsia and different degrees of intrauterine growth restriction.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant danish speeking women

Exclusion Criteria:

* Conditions/diseases involving chronical inflammation, or immunological activity

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women attending nuchal transcluency examination at Gynækologisk-Obstetrisk dept. Roskilde University Hospital
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-11 (Estimated); Study Completion 2012-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Estrid Høgdall, PhD leader, Study Director — Dept of Pathology Herlev Hospital, Denmark; Julia S. Johansen, Dr med prof, Study Director — Dept. of oncology and medicine, Herlev Hospital, Denmark
Locations (1):
- Gynækologisk-Obstetrisk Afdeling, Sygehus Nord, Roskilde, Region Sjælland, Denmark

REFERENCES:
- [Derived] Gybel-Brask D, Hogdall E, Johansen J, Christensen IJ, Skibsted L. Serum YKL-40 and uterine artery Doppler -- a prospective cohort study, with focus on preeclampsia and small-for-gestational-age. Acta Obstet Gynecol Scand. 2014 Aug;93(8):817-24. doi: 10.1111/aogs.12432. Epub 2014 Jun 20. PMID 24861484